CLINICAL TRIAL: NCT01187797
Title: Evaluation of the Effects of a Body-centered Emotional Stimulation in Healthy Persons
Brief Title: Effects of Emotional Stimulation on the Stress Levels of Healthy Persons
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Fernando Dimeo, Charie Universitätsmedizin Berlin
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EA408109
Record Dates: First submitted 2010-08-09; First posted 2010-08-24 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-08

CONDITIONS: Depression; Somatization Disorder; Anger; Anxiety
MeSH Terms: conditions — Depression; Somatoform Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Emotional stimulation

INTERVENTIONS:
Other: Emotional stimulation — Increase of the physical correlates of an emotion

SUMMARY:
The purpose of this study is to evaluate the effects of a short-term emotional stimulation on the mood of healthy persons.

DETAILED DESCRIPTION:
The trial assesses the effects of a emotion-centered stimulation on the mood of healthy persons. The outcomes will be evaluated with standard questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45
* Ability to speak German

Exclusion Criteria:

* Physical or psychiatric disorders
* Consume of drugs or alcohol 24 previous to the test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Depression | After 10 days
  Depression scores will be evaluated with the BDI
Somatization | After 10 days
  Somatization will be assessed with the SOMS7 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany